CLINICAL TRIAL: NCT02240550
Title: A Prospective, Randomized, Double-armed, Single-blinded, Comparative Clinical Study to Evaluate the Effectiveness of ProFlor vs. Lichtenstein for Inguinal Hernia Repair
Brief Title: A Comparative Clinical Study to Evaluate the Effectiveness of ProFlor vs. Lichtenstein for Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insightra Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P0133
Record Dates: First submitted 2014-09-08; First posted 2014-09-15 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Inguinal Hernia
Keywords: Open Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ProFlor Hernia Repair System (Active Comparator): A 3-D hernia mesh
  Interventions: Device: ProFlor Hernia Repair System
- Lichtenstein Hernia Repair (Active Comparator): Using flat polypropylene mesh
  Interventions: Device: Lichtenstein hernia repair

INTERVENTIONS:
Device: ProFlor Hernia Repair System — The 3-D hernia mesh will be used in the repair of your inguinal hernia.
  Other Names: 3D mesh
  Arms: ProFlor Hernia Repair System
Device: Lichtenstein hernia repair — The standard Lichtenstein hernia repair with flat mesh will be used in the treatment of your inguinal hernia.
  Other Names: Polypropylene
  Arms: Lichtenstein Hernia Repair

SUMMARY:
This investigation will be a double-armed, randomized (Blinded patients and Blinded examiner) prospective study designed to collect perioperative and postoperative data to compare the QOL of ProFlor vs. Lichtenstein inguinal hernia repair.

DETAILED DESCRIPTION:
The primary objectives of this study will be to evaluate the immediate and short-term amount of post-operative pain, the quality of life (QOL), as well as return to normal activities (work) for the two procedures. Carolinas Comfort Scale (CCS) and Visual Analogue Score (VAS) assessments will be held at regular intervals to evaluate these objectives.

The secondary objective of the study is to identify any short-term study related complications/adverse events.

The follow up will be immediately post-operative, post-operative day 1, and 1, 2,and 4 weeks. The first and 4th week's visits are mandatory office visits (if possible). If not available for office visit, a CCS assessment will be mailed or will be conducted via phone.

Up to 50 patients may be enrolled for this study (25 per arm). A report may be generated for presentation at an international meeting such as the AHS, EHS, or APHS if decided by the lead investigator.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo routine inguinal hernia repair
* Male and Female patients between 18 and 65 years old
* Competent to give consent
* Clinically relevant inguinal hernia (classification: EHS P L/M 1/2/3)
* Defect size at operation is between 5mm and 35mm
* Diagnosed with unilateral, direct, indirect or mixed inguinal hernia
* Primary hernia at the operative site

Exclusion Criteria:

* Signs of obvious local or systemic infection
* Any previous surgery on the hernia operative site
* Hernia is not in the inguinal area
* Hernia is not identified as indirect or direct
* Femoral hernias
* Known collagen disorder
* Presenting with unstable angina or NYHA class of IV
* Known Pregnancy or Nursing women
* Active drug user
* Recurrence of a repair by any method
* Patients with giant inguinoscrotal hernia or abdominal wall defect >35 mm in diameter - e.g. large direct or combined inguinal hernia type Nyhus IIIb / EHS P L/M 1/2/3
* Immunosuppression, prednisone>15 mg/day, active chemotherapy
* End stage renal disease
* Abdominal ascites
* Skin infection in area of surgical field
* BMI >35
* Peritoneum cannot be closed
* Patient has a clinically relevant co-morbidity (antithrombic prophylaxis due to cardiovascular pathologies, diabetes requiring insulin therapy or immunodeficiency syndrome of any type)
* Neutropenia with absolute neutrophil count (ANC)<500 cells/mm3
* Significant of life-threatening condition (e.g., endocarditis) that would confound or interfere with the procedure
* Patients that require anticoagulant monitoring with an activated partial thromboplastin time (aPTT)
* Patients unwilling to forego blood and/or blood product donation for at least 3 months from initiation of first study device
* Treatment with investigational medicinal product within 30 days before enrollment and for the duration of the study
* Investigational device present, or removed within 30 days before enrollment, or presence of device-related infection
* Patients who the investigator considers unlikely to adhere to the protocol or complete the clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the immediate and short-term amount of pain. | 1 month
  We will evaluate the immediate and short-term amount of pain using the VAS and Carolinas Comfort Scale (CCS) assessments held at regular intervals.
Compare the time required for return to normal activities (work). | 1 month
  We will capture the time required to return to normal activities as indicated by the patient.

SECONDARY OUTCOMES:
Identify any short-term related complication/adverse events associated with the procedures. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: John Murphy, MD, Principal Investigator — Healing Hands Clinic
Locations (1):
- Healing Hands Clinic, Pune, India